CLINICAL TRIAL: NCT02634541
Title: The Efficacy of Adalimumab and Conventional Antirheumatic Drugs in Alleviating Axial and Aortic Inflammation Detected in PET/CT in Patients With Axial Spondyloarthritis
Brief Title: Adalimumab in Alleviating Inflammation in Patients With Axial Spondyloarthritis
Acronym: PETSPA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Helsinki (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Tuomo Nieminen, Professor of Internal Medicine, University of Helsinki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PETSPA; 2015-000752-20 (EudraCT Number)
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Ankylosing Spondyloarthritis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DMARD-naive (Active Comparator): Sulfasalazine will be given as the initial therapy.
  Interventions: Other: PET/CT imaging
- Post-sulfasalazine (Experimental): Sulfasalazine contraindicated or not efficient, adalimumab will be given as the initial therapy.
  Interventions: Drug: Adalimumab; Other: PET/CT imaging

INTERVENTIONS:
Drug: Adalimumab — Biologic drug
  Arms: Post-sulfasalazine
Other: PET/CT imaging — PET/CT imaging

SUMMARY:
Axial spondyloarthritis is an inflammatory rheumatic disease mainly affecting joints in the spine and the sacroiliac joints. Inflammatory pathways are likely the central link from axial spondyloarthritis to the known increased risk of atherosclerotic morbidity. Positron emission tomography (PET) is the most sensitive method to detect inflammatory foci in clinical practice. A few small studies have demonstrated that PET imaging together with computed tomography (PET/CT) detects inflamed tissues in relevant patient groups. One study suggested that antirheumatic treatment diminishes the inflammation detected in PET/CT. No study so far has disclosed whether aortic inflammation is present in patients with spondyloarthritis, and whether the inflammation would wane with efficient antirheumatic treatment. The current study is aimed to grade the articular and aortic inflammatory signals in the PET/CT imaging before and after antirheumatic treatment of clinically active axial spondyloarthritis.

Sixty patients aged 18-75 years with axial spondyloarthritis and radiologic sacroiliitis as detected either by MRI or X-ray will be recruited. Twenty of those are DMARD-naive, and 40 patients have axial spondyloarthritis resistant to sulfasalazine or other conventional antirheumatic drug. In addition, approximately 30 patients without spondyloarthritis but with stable coronary heart disease and approximately 20 healthy controls will be taken as historical controls. All the axial spondyloarthritis patients are PET/CT scanned after inclusion in the study. The DMARD-naive patients (n=20) are started sulfasalazine-based regimen for 12 weeks, which is the time point for a second PET scan for this subgroup. Adalimumab will be commenced for those without remission at 12 weeks. After another 16 weeks, those with adalimumab will be scanned with PET/CT for the third time. The subgroup with active disease in spite of prior conventional treatment (n=40) is also scanned with PET/CT right after the enrolment and after 16-week treatment with adalimumab. The first 15 patients form a pilot group, which is used to check the validity of the power calculation.

The project will give essential new information on PET-detectable inflammation in the patients with axial spondyloarthritis. The results will be published in international publication series. The publications will form the basis for a doctoral thesis. Funding for the project comes from Abbvie Ltd.

ELIGIBILITY:
Inclusion Criteria:

* Axial spondyloarthritis (ASAS criteria) and radiologic sacroiliitis as detected either by MRI or X-ray.

Exclusion Criteria:

* Psoriasis or psoriasis arthropathy
* Inflammatory bowel disease
* Unwillingness to participate in the study with additional imaging protocols
* Expected life-span less than <1 year
* Diabetes (to improve the PET imaging quality)
* Probable noncompliance
* Pregnancy
* Age <18 years or >75 years
* Contraindication for adalimumab
* Methotrexate used within the previous 6 months
* A biologic medicine used within the previous 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
PET signals within groups | 16 weeks
  Decrease in PET signal levels both in major CV tissues (mean TBR in the whole aorta) and musculoskeletal tissues (lumbar spine and articular enthesitis as well as arthritis) after antirheumatic treatment. Thus the variables of most interest reflect intraindividual changes.

SECONDARY OUTCOMES:
PET signals between groups | 16 weeks
  Comparison of the pre-treatment PET signals between the three groups: those with axial spondyloarthritis, historical healthy controls and the patients with coronary heart disease.

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Päijät-Häme Central Hospital, Lahti

IPD SHARING:
Plan to Share IPD: No